CLINICAL TRIAL: NCT02918851
Title: VO2 Max: In Vivo Model for Functional Red Cell Testing. Can RECESS be Explained?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Elliott Bennett-Guerrero, Professor and Vice Chairman, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 953865
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 7-day old RBCs (Experimental): Transfusion of 7-day stored red blood cells: Subjects will be transfused with their own 7-day old red blood cells
  Interventions: Biological: Transfusion of 7-day stored red blood cells
- 28-day old RBCs (Experimental): Transfusion of 28-day stored red blood cells: Subjects will be transfused with their own 28-day old red blood cells
  Interventions: Biological: Transfusion of 28-day stored red blood cells
- 42-day old RBCs (Experimental): Transfusion of 42-day stored red blood cells: Subjects will be transfused with their own 42-day old red blood cells
  Interventions: Biological: Transfusion of 42-day stored red blood cells

INTERVENTIONS:
Biological: Transfusion of 7-day stored red blood cells — Subjects will donate blood at Week 0 and Week 5 of their participation and receive, at Week 6, back a transfusion of their Week 5 (7-day old) red blood cells.
  Arms: 7-day old RBCs
Biological: Transfusion of 28-day stored red blood cells — Subjects will donate blood at Week 2 and Week 5 of their participation and receive, at Week 6, back a transfusion of their Week 2 (28-day old) red blood cells.
  Arms: 28-day old RBCs
Biological: Transfusion of 42-day stored red blood cells — Subjects will donate blood at Week 0 and Week 5 of their participation and receive, at Week 6, back a transfusion of their Week0 (42-day old) red blood cells.
  Arms: 42-day old RBCs

SUMMARY:
This is a single-center, randomized, partially blinded study to determine whether 42-day old red blood cells (RBCs) deliver oxygen as effectively as 7-day old RBCs and also to determine whether transfusion with 28-day old RBCs is non-inferior to 7-day old RBCs with respect to oxygen delivery.

In this study, subjects will be randomized to be transfused with 2 units of autologous (one's own) RBCs that are either 7-, 28-, or 42-days old. Endpoints include changes in exercise duration and VO2 max (test of oxygen consumption/delivery) between groups.

DETAILED DESCRIPTION:
The US Food and Drug Administration (FDA) regulations permit additive-containing RBCs to be stored for up to 42 days prior to transfusion. However, RBCs progressively develop abnormalities during storage. The efficacy of older stored blood, i.e., effective oxygen delivery, has not been established in rigorous controlled studies. Due to pragmatic reasons, a large clinical trial that randomizes patients to "old" blood may not be feasible.

Every subject will have 2 phlebotomy visits at Stony Brook University Hospital. Subjects randomized to the 7- and 42-day old groups will have 2 units of blood removed at Week 0 and another 2 units removed at Week 5. However, the remaining 28-day group will have 2 units of blood removed at Week 2 and only 1 unit of blood removed at Week 5. During week 6, each subjects will have 3 study visits: 1) On Monday, a VO2 max test; 2) On Wednesday, a transfusion with 2 units of autologous RBCs (each over 1 hour), followed by a VO2 max test 2 hours later; 3) On Friday, a VO2 max test will be done in order to calculate a delta VO2 max (Friday minus Monday results).

ELIGIBILITY:
Inclusion Criteria:

* Habitual exerciser defined as ≥ 30 minutes of at least moderate or high intensity exercise ≥ 3 times per week. After consent, and at the subsequent screening visit, a VO2 max test will be performed, and subjects with a low value (< 35 mL/kg/min) will be excluded (screen failure). Based on our previous experience, we anticipate that <10% of the subjects will fall into this category
* Calculated total blood volume (TBV) ≥4,500 mL using an established formula:

  1. Men: (0.006012 x H3) + (14.6 x W) + 604 = TBV
  2. Women: (0.005835 x H3) + (15 x W) + 183 = TBV [H=height in inches; W=weight in pounds]
* Has access to transportation to visit the blood collection facility and to return to Stony Brook for all study visits.

Exclusion Criteria:

* Any significant acute or chronic medical illness or problem, including, but not limited to, diabetes, hypertension, cardiac disease, asthma, chronic obstructive lung disease
* Current or recent (last 60 days) tobacco or nicotine use
* History of sickle cell trait or disease or any other acquired or hereditary hematological abnormality
* History of fainting or other significant adverse reaction during phlebotomy or donation of blood
* Known prolonged corrected QT interval (or evidence of such at screening) on electrocardiogram defined as >470 ms
* Known or suspected illicit drug or alcohol abuse
* Known or suspected HIV, Hepatitis B, or Hepatitis C infection
* History of thrombophilia or anticoagulant therapy
* Pregnancy
* Obesity defined as BMI>30
* Recent history of blood donation: a) Single whole blood unit donation within the past 8 weeks; b) Double RBC donation by apheresis within the past 16 weeks; or c) Plasma donation by apheresis within the past 4 weeks
* Inadequate RBC mass based on TBV <4500 ml (above) or screening Hb <14 g/dL

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Bennett-Guerrero, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook Medicine, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bennett-Guerrero E, Rizwan S, Rozensky R, Romeiser JL, Brittelli J, Makaryus R, Lin J, Galanakis DK, Triulzi DJ, Moon RE. Randomized controlled trial of 7, 28, vs 42 day stored red blood cell transfusion on oxygen delivery (VO2 max) and exercise duration. Transfusion. 2021 Mar;61(3):699-707. doi: 10.1111/trf.16237. Epub 2020 Dec 27. PMID 33368319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 randomized
Period: Overall Study
Arm/Group | 7-day Old RBCs | 28-day Old RBCs | 42-day Old RBCs
Started | 14 | 14 | 14
Completed | 10 | 10 | 10
Not Completed | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7-day Old RBCs | 28-day Old RBCs | 42-day Old RBCs | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22.5 [20 to 25] | 23.5 [22 to 25] | 23 [22 to 27] | 23 [22 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 9 | 8 | 10 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 6 | 6 | 5 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Maximal Oxygen Uptake (VO2 Max) After Blood Cell Transfusion
Description: Percent Change From Baseline in Maximal Oxygen Uptake (VO2 Max) on Day 2 After Blood Cell Transfusion
Time Frame: Baseline (prior to receiving blood) and Day 2 after receiving blood
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | 7-day Old RBCs | 28-day Old RBCs | 42-day Old RBCs
Number analyzed (Participants) | 10 | 10 | 10
percent change | 10.5 [0.2 to 17.3] | 8.5 [2.9 to 13.1] | 10.9 [5.7 to 16.8]

2. Secondary Outcome: Percent Change in Duration of Exercise From Baseline to Day 2 After RBC Transfusion
Description: Percent change in duration of exercise from baseline to day 2 after red blood cell transfusion
Time Frame: Baseline and Day 2 after transfusion
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | 7-day Old RBCs | 28-day Old RBCs | 42-day Old RBCs
Number analyzed (Participants) | 10 | 10 | 10
percent change | 5.4 [4.1 to 6.9] | 5.4 [0.2 to 9.2] | 4.9 [2.0 to 7.2]

ADVERSE EVENTS:
Time Frame: End of study an average of 2 months
Arm/Group | 7-day Old RBCs | 28-day Old RBCs | 42-day Old RBCs
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02918851/Prot_SAP_000.pdf